CLINICAL TRIAL: NCT01017302
Title: A Randomized, Double-blind, Placebo-controlled, Titration Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Dose and Escalating Doses of RO5095932 in Patients With Type 2 Diabetes Mellitus on Stable Background Therapy
Brief Title: A Study With RO5095932 in Patients With Type 2 Diabetes on Stable Metformin Therapy.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NP22709
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: RO5095932
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 3 (Experimental)
  Interventions: Drug: RO5095932
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Subcutenaous once weekly for 4 weeks
  Arms: 2
Drug: Placebo — Single subcutaneous dose in week 5
  Arms: 4
Drug: RO5095932 — Escalating subcutaneous doses once weekly over a 4 weeks period
  Arms: 1
Drug: RO5095932 — Single subcutenaous dose in week 5
  Arms: 3

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of RO5095932 in adult patients with type 2 diabetes mellitus. Patients that are on stable metformin therapy are eligible to enter the study. There will be a 5-weeks exenatide run in period and a 5-weeks period when co-administered with the study drug. RO5095932 will be administered subcutaneously as a single dose or as escalating doses. Patients will be randomized to receive either active drug or placebo in weeks 1 to 4. Active drug or placebo will be administered once weekly for 4 weeks. Patients who received active drug in weeks 1 to 4 will receive placebo in week 5. Patients who received a single dose of placebo in weeks 1 to 4, will receive a single dose of active drug in week 5. The anticipated time of study treatment is <6 months. The target sample size is <100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-65 years of age
* Diabetes mellitus, type 2 for at least 6 months before screening
* On treatment with stable doses of metformin for at least 3 months before screening
* BMI between >/=25 and </=39

Exclusion Criteria:

* Type 1 diabetes
* Pancreatitis
* Treatment with insulin for more than one week within 3 months prior to study start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of various doses of RO5095932 | Weeks 1-4, 6, 8

SECONDARY OUTCOMES:
Safety and Tolerability of a single dose of RO5095932 | Week 5, 6, 8
Pharmacokinetics: blood concentration | Weeks 1-4, 6, 8
Pharmacodynamics: glucose, insulin, C-peptide | Weeks 1-4, 6, 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- San Antonio, Texas, United States